CLINICAL TRIAL: NCT00372242
Title: Feasible Means to Address Moderately Malnourished Children Within BINP Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 99-041
Record Dates: First submitted 2006-09-04; First posted 2006-09-06 (Estimated); Last update posted 2006-09-06 (Estimated); Status verified 2003-04

CONDITIONS: Mild and Moderate Malnourished Children
Keywords: Mal-nutrition; Morbidity; Nutrition Education; Complementary Feeding; Weight gain; Height
MeSH Terms: conditions — Lymphoma, Follicular; Weight Gain

INTERVENTIONS:
Behavioral: Prospective Longitudinal Interventional Stury

SUMMARY:
The Bangladesh Integrated Nutrition Project (BINP) of the Government of Bangladesh has started showing reduction in malnutrition of women and children under two years of age in last 3 years of it's activities. That was a demonstration study to test the efficacy of the approach on a relatively small number of children with intensive intervention. A study will be therefore conducted in 4 division of BINP thanas of Bangladesh over an 18-month period. Moderately malnourished children will be in management intervention and mildly malnourished and well-nourished infants will be in preventive intervention group. For management intervention, a total of 750 moderately malnourished will be randomized to receive either intensive nutrition education or less intensive education. For preventive purpose, 380 mildly malnourished children of 6 months to 2 years of age and 240 well nourished infants of 6 to 9 months of age will receive either less intensive education or no education. Infants between 6 to 9 month ages will be brought under less INE to ensure their complementary feeding practice. Care givers of one group of mildly malnourished children and one group of 6-9 month old infants will not receive any education to serve as controls. Focus group discussion will be held before the educational intervention to identify the perception of the mother, her husband and female decision maker of her family on child nutrition, caring practice and common practice of health care. BCC materials will be developed after FGD and that will be used during nutrition education. Mothers of the first intervention group will receive intensive nutrition education for child feeding twice weekly for first three months, which will be then reinforced once in a week for the last three months of intervention. The less intensive intervention group will receive nutrition education twice a week for the first month then once a week for two months and then twice monthly for the last three months of intervention. INE will be given for a total of 6 months. An observation will be done to identify for sustainability effect for an additional period of 6 months. Their weight and length gain will be recorded. It is expected that the results of the study will help define the effectiveness of our nutrition education package to prevent and reduce moderate malnutrition existing in large proportion of children in setting with different geographical, and cultural and feeding practices.

DETAILED DESCRIPTION:
Bangladesh has the highest proportion of malnourished children in the world. The infant and child mortality are also among the highest in south Asia. In Bangladesh, '. The Government of Bangladesh has been trying different ways for reducing childhood malnutrition. Such programs include the Vulnerable Group Development (VGD) Project, vitamin A distribution project, iodine deficiency disorder control program, iron supplementation program and improving food availability for the underprivileged sections of the society. Despite these, not enough improvement has been observed in the field of nutrition. In review of the past fifty-year's information of dietary intake and growth, it has been observed that food intake has substantially decreased and growth faltering in children has worsened (Roy et al 1988). Materal malnutrition is evidenced by low weight, short stature and anemia in pregnant and lactating women. Micronutrient deficiencies are evidenced by prevalence of xerophthalmia, iron deficiency anemia and iodine deficiency disorders. The effects of childhood under nutrition, begin with a low birth weight (estimated to occur among 35-50% of births in Bangladesh) (Hasan et al 1995) and continue into adulthood.

The prevalence of PEM among children is very high, and has remained almost the same for the last decade. Thirty percent of all children under six years of age are severely stunted and another 31.2% are moderately stunted (BBS 1995). As many as 68.3% of the total children are under -weight and 16.7% are wasted, the highest rates are in Asia (BBS 1995). Given the greatly disadvantaged start by the way of a low birth-weight followed by inadequate breast-feeding by their undernourished mothers, average Bangladeshi infants are already below the lower end of the range of anthropometric values found among western babies during the first three to six months. The late and insufficient introduction of complementary feeding further retards the infant's growth; usually the child do not pick up its pace of growth before two years of age. By then, it is too late to reverse the early growth lag, which persists throughout the life, and similarly some of the damages done to mental development are irreparable. The weight for age curve of Bangladeshi children continues to lie below the third percentile of the NCHS Standard, though it runs roughly parallel to the standard from around the second year of life onward; the older children cope better with the adverse milieu of food-insecure and unhealthy household, while being unable to regain lost ground.

ELIGIBILITY:
Inclusion Criteria:

* Mildly malnourished children without growth faltering aged 6 to 24 months
* Moderately malnourished children without growth faltering aged 6 to 24 months
* Well-nourished children aged 6 to 9 months

Exclusion Criteria:

* >2 years children
* Severely malnourished children

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1231
Dates: Start 2000-12; Study Completion 2002-09

PRIMARY OUTCOMES:
Mothers understanding and ability to identify moderate malnutrition in children.
Mothers understanding on consequence of moderate malnutrition.
Change in knowledge of mothers in feeding practices.
Frequency of home feeding (Breast-feeding and supplementary feeding).
Frequency of seeking medical care during illness, referral, incidence, duration of illness.
Adequacy of child feeding, frequency & type of feeding.
Weight gain, weight for age and weight for height at the end of intervention.
Proportion of complementary feeds in 6-9 months age group.
Nutritional status of children at various phases of intervention and observation.
Adaptation level of nutrition education program by CNP, CNO.
Constant of not practicing education knowledge.

SECONDARY OUTCOMES:
Incidence and prevalence of diarrhoea and ALRI
Referral success and failure
Resistance to education
Food insecurity for child
Mothers time constraint for CF preparation
CNP time constraints for INE

CONTACTS AND LOCATIONS:
Overall Officials: Swapan K Roy, MBBS, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh